CLINICAL TRIAL: NCT00261963
Title: The Effect of UV-Irradiation on Cutaneous Cicatrices -A Randomised, Controlled Study With Clinical, Skin Reflectance, Histological and Biochemical Evaluations
Brief Title: The Effect of UV-Irradiation on Cutaneous Cicatrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: KF 01-187-03
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Skin Cicatrices

INTERVENTIONS:
Device: ultraviolet light

SUMMARY:
The purpose of this study is to examine the effect of UV-irradiation on human cutaneous cicatrices by clinical examinations and histological, immunohistochemical and biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking volunteers,
* Skintypes II or III

Exclusion Criteria:

* Atopic dermatitis,
* Tendency to produce keloids or hypertrophic scars,
* Exposure of UV light during the last 3 months,
* Medical treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2004-02; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Eva Due, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark